CLINICAL TRIAL: NCT01973439
Title: PENTA15: Plasma Pharmacokinetic Study of Once Versus Twice Daily Abacavir as Part of Combination Antiretroviral Therapy in Children With HIV-1 Infection Aged 3 Months to <36 Months
Brief Title: PENTA15: Pharmacokinetic Study of Once Versus Twice Daily Abacavir in HIV-1 Infected Children Aged 3 to <36 Months
Acronym: PENTA15
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PENTA15; 2005-004433-18 (EudraCT Number)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infection
Keywords: HIV; Abacavir; Lamivudine; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abacavir Once versus Twice Daily (Other): This is a single arm study. Intervention 1: PK assessment while on Twice Daily Abacavir (Week 0) Intervention 2: PK assessment while on Once Daily Abacavir (Week 4)
  Interventions: Other: Intervention 1: PK assessment while on Twice Daily Abacavir; Other: Intervention 2: PK assessment while on Once Daily Abacavir

INTERVENTIONS:
Other: Intervention 1: PK assessment while on Twice Daily Abacavir — Week 0
  Other Names: Ziagen; ABC
Other: Intervention 2: PK assessment while on Once Daily Abacavir — Week 4
  Other Names: Ziagen; ABC

SUMMARY:
To compare the plasma pharmacokinetic (PK) parameters of q24h versus q12h dosing of abacavir in HIV-1-infected infants and children aged 3 months to 36 months

The secondary objectives of PENTA15 were:

To compare the plasma PK parameters of q24h versus q12h dosing of lamivudine in HIV-1-infected infants and children aged 3 months to 36 months who were receiving lamivudine in combination with abacavir

To compare age-related differences in the PK parameters of q24h versus q12h dosing of abacavir and lamivudine infants and children in 3 age groups (≥3 to <12 months, ≥12 to <24 months and ≥24 to <36 months)

To describe child and family acceptability of and adherence to q24h compared to q12h dosage regimens of abacavir and lamivudine

ELIGIBILITY:
Inclusion Criteria:

* Infants and children with confirmed presence of HIV-1 infection
* Infants and children aged 3 to <36 months
* Parents/guardians able and willing to give written, informed consent
* Currently on combination ART including Abacavir (ABC) oral solution with or without Lamivudine (3TC) oral solution, for at least 12 weeks and expected to stay on this regimen for at least a further 12 weeks.
* HIV-1 RNA viral load either;

  * suppressed HIV-1 RNA viral load (i.e. <400 copies/ml)
  * non-suppressed, but low, HIV-1 RNA viral load (i.e. 400-20 000 copies/ml). The non-suppressed children should have had a stable or decreasing HIV-1 RNA viral load prior to study entry and should be considered to be still gaining benefit from the current regimen
* Stable or rising CD4+ cell percent prior to study entry and should not be expected to fall within the next 12 weeks.

Exclusion Criteria:

* Intercurrent illness
* Receiving concomitant therapy except prophylactic antibiotics
* Abnormal renal or liver function (grade 3 or above)

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- France (2):
  - Hôpital Port Royal, Paris
  - Hôpital Robert Debré, Paris
- Immundefekt-Ambulanz, Dr. von Haunersches Kinderspital, Munich, Germany
- Clinica Pediatrica, Università di Padova, Padua, Italy
- Spain (3):
  - Hospital Universitario, Getafe
  - Hospital 12 de Octubre, Madrid
  - Hospital Gregorio Maranon, Madrid
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Evelina Children's Hospital, London
  - St. Mary's Hospital, London

REFERENCES:
- [Background] Paediatric European Network for Treatment of AIDS (PENTA). Pharmacokinetic study of once-daily versus twice-daily abacavir and lamivudine in HIV type-1-infected children aged 3-<36 months. Antivir Ther. 2010;15(3):297-305. doi: 10.3851/IMP1532. PMID 20516550

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: This is a single arm crossover study
  1. st intervention: PK assessment while on Twice Daily Abacavir
  2. nd intervention: PK assessment while on Once Daily Abacavir
Period: Overall Study
Arm/Group | Single Arm
Started | 23
Two Evaluable PK Days | 18 (18 Children had two evaluable PK days)
One Evaluable PK Day Only | 5 (5 children had only one evaluable PK day.)
Completed | 18
Not Completed | 5
Not completed — Lost samples from one PK Day | 2
Not completed — Vomiting after commencing once daily | 1
Not completed — PK curve incomplete | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: This is a single arm crossover study First intervention: PK assessment while on Twice Daily Abacavir Second intervention: PK assessment while on Once Daily Abacavir
Arm/Group | Single Arm
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3
  Black, African or other | 14
  Mixed Black/White | 1
Region of Enrollment [Number; unit: participants]
  Germany | 3
  Italy | 1
  United Kingdom | 9
  Spain | 2
  France | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) (0-24) of Abacavir on Twice Daily Dosing
Description: Blood samples were taken at 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 12 hours post-ingestion of medication.
Time Frame: Week 0
Measure: Geometric Mean (95% Confidence Interval); unit: h*mg/L
Groups:
- Single Arm: This is a single arm study. First intervention: PK assessment of Twice Daily Abacavir (Week 0) Second intervention: PK assessment of Once Daily Abacavir (Week 4)
Arm/Group | Single Arm
Number analyzed (Participants) | 18
h*mg/L | 10.85 [8.89 to 13.24]

2. Primary Outcome: Cmax of Abacavir on Twice Daily Dosing
Description: Blood samples were taken at 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 12 hours post-ingestion of medication.
Time Frame: Week 0
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Single Arm
Number analyzed (Participants) | 18
mg/L | 2.29 [1.80 to 2.91]

3. Primary Outcome: AUC(0-24) of Abacavir on Once Daily Dosing
Description: Blood samples were taken at 0 (pre-dose), 1, 2, 3, 4, 6, 8, 12 and 24 hours post-ingestion of medication
Time Frame: Week 4
Measure: Geometric Mean (95% Confidence Interval); unit: h*mg/L
Arm/Group | Single Arm
Number analyzed (Participants) | 18
h*mg/L | 11.57 [9.89 to 13.53]

4. Primary Outcome: Cmax of Abacavir on Once Daily Dosing
Description: Blood samples were taken at 0 (pre-dose), 1, 2, 3, 4, 6, 8, 12 and 24 hours post-ingestion of medication.
Time Frame: Week 4
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Single Arm
Number analyzed (Participants) | 18
mg/L | 4.68 [3.86 to 5.67]

ADVERSE EVENTS:
Arm/Group | Abacavir Once Versus Twice Daily
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abacavir Once Versus Twice Daily (N=23)
Croup Infectious (Infections and infestations) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Gastroenteritis Bacteria (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less